CLINICAL TRIAL: NCT06063083
Title: Addressing Latino Men Who Have Sex With Men (MSM) Health Disparities by Increasing Engagement With Behavioral and HIV Prevention Services: An Implementation Science Approach
Brief Title: Tell Me More ("Dime Mas")
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Audrey Harkness, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20201189; K23MD015690 (NIH)
Record Dates: First submitted 2023-09-22; First posted 2023-10-02 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: HIV; Mental Health Issue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tell Me More ("Dime Mas") group (Experimental): Participants will get the Tell Me More ("Dime Mas") program within up to 6 months.
  Interventions: Behavioral: Tell Me More ("Dime Mas"); Behavioral: Peer Ambassador Stories [Listen Miami ("Oye Miami")]; Behavioral: Standard Community Outreach
- Peer Ambassador Stories [Listen Miami ("Oye Miami")] group (Experimental): Participants will get the Peer Ambassador Stories [Listen Miami ("Oye Miami")] within up to 6 months.
  Interventions: Behavioral: Peer Ambassador Stories [Listen Miami ("Oye Miami")]; Behavioral: Standard Community Outreach
- Standard Community Outreach group (Active Comparator): Participants will receive standard community outreach within up to 6 months.
  Interventions: Behavioral: Standard Community Outreach

INTERVENTIONS:
Behavioral: Tell Me More ("Dime Mas") — Participants will receive an initial approximately 1 hour outreach session followed by up to 3 approximately monthly check-in outreach attempts (approximately 15 minutes each). All study visits can be done in person or remotely. Each contact will involve helping participants get connected to PrEP, HIV testing, and behavioral health treatment.
  Arms: Tell Me More ("Dime Mas") group
Behavioral: Peer Ambassador Stories [Listen Miami ("Oye Miami")] — Participants will receive a link to a website featuring stories of local Latino MSM using PrEP, HIV testing, and behavioral health treatments. Participants will receive intermittent (based on personal choice) reminders to view the website. The website will also show referrals to services and provide the option to submit a story via written, video, or audio recording. Participants can access the website using a personal electronic device at any time during within the study period.
  Arms: Peer Ambassador Stories [Listen Miami ("Oye Miami")] group; Tell Me More ("Dime Mas") group
Behavioral: Standard Community Outreach — Participants will receive the standard community outreach, which will be a list of referrals for HIV testing, PrEP, and behavioral health treatments.

SUMMARY:
This study will be used to develop a program to help Latino men who have sex with men obtain pre-exposure prophylaxis (PrEP), HIV testing, and behavioral health services. The project will then involve a pilot test of this program with a community partner.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Latino/Hispanic
* identify as a sexual minority man (e.g., gay, bisexual) and/or a man who has sex with men
* age 18 years or older
* English and/or Spanish speaking
* self-report an HIV-negative or unknown HIV status
* currently reside in the greater Miami area
* PrEP eligible (based on Centers for Disease Control (CDC) criteria) and not currently taking PrEP adherently
* self-report experiencing one or more clinically significant behavioral health concerns (mental health, substance use) and/or are not currently receiving behavioral health services or self-report an unmet need for behavioral health services

Exclusion Criteria:

* Unable to provide consent
* Opinion of the PI that the participant would be at risk for harm to self or others
* Have a medical or psychiatric condition that would interfere with ability to participate in study procedures in the opinion of the PI
* Involvement in any other HIV prevention or behavioral health study that may interfere with the ability to test major study outcomes (evaluated by the PI on a case-by-case basis)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as a man
Enrollment: 90 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in PrEP Engagement, as measured by the PrEP cascade questionnaire | Baseline, 3 months, 6 months
  This will be assessed using the PrEP cascade measure, which specified five "levels" of PrEP engagement (i.e., pre-contemplation, contemplation, preparation, action, and maintenance). We will evaluate this outcome as an ordered-categorical outcome.

SECONDARY OUTCOMES:
Change in Behavioral Health Treatment Engagement, as measured by the Behavioral health cascade questionnaire (based on the Psychosocial Treatment Inventory) | Baseline, 3 months, 6 months
  We will use a modified version of the Psychosocial Treatment Inventory to assess participants' engagement with behavioral health treatment (inclusive of mental health or substance use treatment). This measure evaluates five "levels" of behavioral health treatment engagement (i.e., pre-contemplation, contemplation, preparation, action, and maintenance). We will evaluate this outcome as an ordered-categorical outcome.
Change in Recent (within the last 3 months) HIV testing | Baseline, 3 months, 6 months
  Participants will answer a question about being tested in the past three months. A score of 1 means that the participant received at HIV test in the last three months. A score of 0 means the participant did not.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Harkness, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No